CLINICAL TRIAL: NCT01122446
Title: A Double-blind, Randomized Investigator-initiated Study to Determine the Safety and the Effect of Diamyd® on the Progression to Type 1 Diabetes in Children With Multiple Islet Cell Autoantibodies
Brief Title: Diabetes Prevention - Immune Tolerance
Acronym: DIAPREV-IT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, Helena Elding Larsson, MD PhD, Lund University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DIAPREV/2008
Record Dates: First submitted 2010-05-12; First posted 2010-05-13 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Prediabetes; Type 1 Diabetes
Keywords: Alum-GAD; Type 1 diabetes; prevention; immune tolerance; glucose tolerance; glutamate decarboxylase autoantibodies
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo comparator (Placebo Comparator): Two doses of placebo day 1 and 30
  Interventions: Other: Placebo comparator
- Alum-GAD (Diamyd) (Active Comparator): 20 microgram Diamyd day 1 and 30
  Interventions: Drug: Diamyd

INTERVENTIONS:
Other: Placebo comparator — Placebo comparator day 1 and 30 in non-diabetic children with multiple islet autoantibodies.
  Post diagnosis: Two doses of 20 microgram Diamyd day 1 and 30 in children originally receiving placebo.
  Arms: Placebo comparator
Drug: Diamyd — 20 microgram day 1 and 30 in non-diabetic children with multiple islet autoantibodies.
  Post diagnosis: Two doses of Diamyd followed to children originally receiving Diamyd
  Other Names: Alum-GAD
  Arms: Alum-GAD (Diamyd)

SUMMARY:
A double-blind, randomized investigator-initiated study to determine the safety and the effect of Diamyd® on the progression to type 1 diabetes in children with multiple islet cell autoantibodies

Eligible children are 4 years or older, have positive GAD-antibodies and at least one additional autoantibody and not yet diabetes.

Objectives:

DiAPREV-IT is the first prevention study with Diamyd®, where the drug is given before onset of type 1 diabetes.

The primary objective is to demonstrate that Diamyd® is safe in children at risk for type 1 diabetes.

The secondary objective is to evaluate if Diamyd® may delay or stop the autoimmune process leading to clinical type 1 diabetes in children with ongoing persistent beta-cell autoimmunity as indicated by multiple positive islet cell autoantibodies.

DETAILED DESCRIPTION:
A double-blind, randomized investigator-initiated study to determine the safety and the effect of Diamyd® on the progression to type 1 diabetes in children with multiple islet cell autoantibodies

Eligible children are 4 years or older, have positive GAD-antibodies and at least one additional autoantibody and not yet diabetes.

Objectives:

DiAPREV-IT is the first prevention study with Diamyd®, where the drug is given before onset of type 1 diabetes.

The primary objective is to demonstrate that Diamyd® is safe in children at risk for type 1 diabetes.

The secondary objective is to evaluate if Diamyd® may delay or stop the autoimmune process leading to clinical type 1 diabetes in children with ongoing persistent beta-cell autoimmunity as indicated by multiple positive islet cell autoantibodies.

Procedure:

50 children will be randomized to 2 injections of Diamyd® or placebo. In DIAPREV-IT we will use the previously tested dose of 20 µg Diamyd® administered as a prime-and-boost at days 1 and 30, as no serious adverse reactions have been observed with this regimen. The children will be followed every 3rd month for 5 years. Before the first injection of study drug both intravenous (IvGTT) and oral (OGTT) glucose tolerance test will be performed. These will be repeated during the study with OGTT every 6 month visit and IvGTT every full year visit.

Safety variables:

Collection of adverse events, serious adverser events, hematology, chemistry, titles of autoantibodies.

Effect variables:

The cumulative incidence of diabetes onset over time since randomization within each treatment group will be estimated using the Kaplan-Meier method (proportion surviving diabetes-free as a function of time).

Secondary efficacy variables:

Change in first-phase insulin response and K-value on IvGTT from baseline Change in fasting, 120 minutes and AUC C-peptide levels on OGTT Change in fasting, 120 minutes and AUC glucose on OGTT Change in HbA1c from baseline All measures during 5 years follow-up.

Children developing diabetes in the study will be offered to participate in a postdiagnosis protocol. Children who have had two doses of active Diamyd in the main study will be given one additional dose of 20 microgram Diamyd followed by one dose of placebo after 30 days. Children who have had two doses of placebo will be given two doses of 20 microgram Diamyd with 30 days in between. Post diagnosis follow up will proceed for at least 15 months from the first post diagnosis injection with collection of adverse events and metabolic evaluation with Mixed meal tolerance tests.

ELIGIBILITY:
Inclusion Criteria:

1. Children from four (4) years of age and participating in DiPiS, TEDDY or Trial Net.
2. Positive GAD65Ab and at least one additional type 1 diabetes-associated autoantibody (IA-2Ab, ZnT8R/W/QAb or IAA).
3. Written informed consent from the child and the child's parents or legal acceptable representative(s) according to local regulations.

Exclusion Criteria:

1. Ongoing treatment with immunosuppressant therapy (topical or inhaled steroids are accepted).
2. Diabetes.
3. Treatment with any oral or injected anti-diabetic medications.
4. Significantly abnormal hematology results at screening.
5. Clinically significant history of acute reaction to vaccines or other drugs.
6. Treatment with any vaccine, other than influenza, within one month prior to the first dose of the study drug or planned treatment with vaccine up to two months after the last injection with the study drug.
7. A history of epilepsy, serious head trauma or cerebrovascular accident, or clinical features of continuous motor unit activity in proximal muscles.
8. Participation in other clinical trials with a new chemical entity within the previous 3 months.
9. Significant illness other than diabetes within 2 weeks prior to first dosing.
10. Known human deficiency virus (HIV) or hepatitis.
11. Presence of associated serious disease or condition, including active skin infections that preclude subcutaneous injection, which in the opinion of the investigators makes the patient non-eligible for the study.
12. Diabetes-protective HLA-DQ6-genotype.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Elding Larsson, MD, PhD, Principal Investigator — Region Skåne and Lund University
Locations (1):
- Clinical Research Center, Pediatric Endocrinology, Jan Waldenströms gata 35, 60:11, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Andersson C, Carlsson A, Cilio C, Cedervall E, Ivarsson SA, Jonsdottir B, Jonsson B, Larsson K, Neiderud J, Lernmark A, Elding Larsson H; DiAPREV-IT Study Group. Glucose tolerance and beta-cell function in islet autoantibody-positive children recruited to a secondary prevention study. Pediatr Diabetes. 2013 Aug;14(5):341-9. doi: 10.1111/pedi.12023. Epub 2013 Mar 8. PMID 23469940
- [Result] Elding Larsson H, Larsson C, Lernmark A; DiAPREV-IT study group. Baseline heterogeneity in glucose metabolism marks the risk for type 1 diabetes and complicates secondary prevention. Acta Diabetol. 2015 Jun;52(3):473-81. doi: 10.1007/s00592-014-0680-1. Epub 2014 Nov 8. PMID 25381193
- [Result] Elding Larsson H, Lundgren M, Jonsdottir B, Cuthbertson D, Krischer J; DiAPREV-IT Study Group. Safety and efficacy of autoantigen-specific therapy with 2 doses of alum-formulated glutamate decarboxylase in children with multiple islet autoantibodies and risk for type 1 diabetes: A randomized clinical trial. Pediatr Diabetes. 2018 May;19(3):410-419. doi: 10.1111/pedi.12611. Epub 2017 Nov 24. PMID 29171140

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Comparator: Two doses of placebo day 1 and 30
  Placebo comparator: Placebo comparator day 1 and 30 in non-diabetic children with multiple islet autoantibodies.
  Post diagnosis: Two doses of 20 microgram Diamyd day 1 and 30 in children originally receiving placebo.
- Alum-GAD (Diamyd): 20 microgram Diamyd day 1 and 30
  Diamyd: 20 microgram day 1 and 30 in non-diabetic children with multiple islet autoantibodies.
  Post diagnosis: Two doses of Diamyd followed to children originally receiving Diamyd
Period: Overall Study
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd) | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 13 | 14 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Adverse events, serious adverse events, hematology, chemistry, autoantibody titles by treatment group
Time Frame: During 5 years follow up from treatment
Measure: Number; unit: Serious adverse events
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Number analyzed (Participants) | 25 | 25
Serious adverse events | 2 | 2

2. Secondary Outcome: Number of Participants With Type 1 Diabetes
Description: Onset of Type 1 diabetes, defined according to ADA criteria, by treatment
Time Frame: During 5 years follow up from treatment
Population: Number of participants developing diabetes during 5 year follow up in each group
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Number analyzed (Participants) | 25 | 25
Participants | 10 | 8

3. Secondary Outcome: Fasting Glucose Over Time
Description: Fasting glucose is measured at baseline and every 6 months within the study. Glucose is analysed by Hemocue.
Time Frame: During 5 year follow-up from treatment
Population: Children meeting the primary endpoint type 1 diabetes are not included in the analysis - therefore the number of analysed children drops during follow-up.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Number analyzed (Participants) | 25 | 25
mmol/L
  0 months | 4.67 (0.56) | 4.74 (0.49)
  6 months: number analyzed (Participants) | 24 | 25
  6 months | 4.98 (0.77) | 5.04 (0.60)
  18 months: number analyzed (Participants) | 23 | 23
  18 months | 5.23 (1.65) | 4.87 (0.71)
  30 months: number analyzed (Participants) | 21 | 20
  30 months | 5.10 (0.61) | 5.05 (0.68)
  42 months: number analyzed (Participants) | 16 | 19
  42 months | 5.13 (0.66) | 4.88 (0.71)
  54 months: number analyzed (Participants) | 15 | 17
  54 months | 5.29 (0.50) | 5.36 (0.39)

4. Secondary Outcome: 120 Minutes Glucose From OGTT Over Time
Description: OGTT is performed at baseline, after 6 months and thereafter annually. Children meeting the primary endpoint type 1 diabetes are not included in the analysis - therefore the number of analysed children drops during follow-up.
Time Frame: During 5 year follow-up from treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol//L
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Number analyzed (Participants) | 24 | 25
mmol//L
  0 months | 6.88 (1.61) | 6.82 (2.12)
  6 months | 7.00 (1.86) | 7.30 (1.87)
  18 months: number analyzed (Participants) | 22 | 23
  18 months | 7.19 (2.05) | 6.41 (1.85)
  30 months: number analyzed (Participants) | 21 | 20
  30 months | 6.54 (1.38) | 6.31 (1.65)
  42 months: number analyzed (Participants) | 16 | 19
  42 months | 6.63 (2.41) | 6.54 (1.30)
  54 months: number analyzed (Participants) | 15 | 17
  54 months | 6.67 (2.38) | 7.04 (3.11)

5. Secondary Outcome: AUC Glucose From OGTT Over Time
Description: OGTT is performed at baseline, after 6 months and thereafter annually.
Time Frame: During 5 year follow-up from treatment
Population: Children meeting the primary endpoint type 1 diabetes are not included in the analysis - therefore the number of analysed children drops during follow-up. One child did not do OGTT at baseline and therefore the placebo group only contains 24 participants in this analysis. At 42 months one additional child only did 2 point OGTT.
Measure: Mean (Standard Deviation); unit: mmol*min/L
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Number analyzed (Participants) | 24 | 25
mmol*min/L
  0 months | 989.63 (207.07) | 938.72 (190.87)
  6 months: number analyzed (Participants) | 23 | 24
  6 months | 973.48 (188.48) | 960.04 (182.05)
  18 months: number analyzed (Participants) | 22 | 21
  18 months | 1005.0 (234.99) | 904.71 (210.34)
  30 months: number analyzed (Participants) | 21 | 19
  30 months | 970.81 (198.96) | 946.16 (175.60)
  42 months: number analyzed (Participants) | 14 | 17
  42 months | 965.43 (323.95) | 967.41 (131.75)
  54 months: number analyzed (Participants) | 15 | 17
  54 months | 949.20 (263.67) | 994.88 (229.35)

6. Secondary Outcome: Fasting C-peptide Over Time
Description: Fasting C-peptide is performed at baseline and thereafter every 6 months
Time Frame: During 5 year follow-up from treatment
Population: Children meeting the primary endpoint type 1 diabetes are not included in the analysis - therefore the number of analysed children drops during follow-up. At 42 months one value is missing due to missed sampling.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Number analyzed (Participants) | 25 | 25
nmol/L
  0 months | 0.18 (0.09) | 0.21 (0.10)
  6 months: number analyzed (Participants) | 23 | 24
  6 months | 0.21 (0.17) | 0.26 (0.10)
  18 months: number analyzed (Participants) | 22 | 22
  18 months | 0.27 (0.18) | 0.30 (0.13)
  30 months: number analyzed (Participants) | 21 | 19
  30 months | 0.34 (0.14) | 0.39 (0.20)
  42 months: number analyzed (Participants) | 14 | 16
  42 months | 0.37 (0.17) | 0.40 (0.23)
  54 months: number analyzed (Participants) | 15 | 16
  54 months | 0.48 (0.25) | 0.45 (0.16)

7. Secondary Outcome: 120 Min C-peptide on OGTT Over Time
Description: OGTT is performed at baseline, after 6 months and thereafter annually
Time Frame: During 5 year follow-up from treatment
Population: Children meeting the primary endpoint type 1 diabetes are not included in the analysis - therefore the number of analysed children drops during follow-up. 120 min C-peptide missing at some endpoints due to missed sample
Measure: Mean (Standard Deviation); unit: nmol//L
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Number analyzed (Participants) | 24 | 25
nmol//L
  0 months | 1.09 (0.60) | 1.22 (0.46)
  6 months: number analyzed (Participants) | 23 | 25
  6 months | 1.04 (0.41) | 1.31 (0.50)
  18 months: number analyzed (Participants) | 22 | 22
  18 months | 1.27 (0.33) | 1.25 (0.39)
  30 months: number analyzed (Participants) | 21 | 20
  30 months | 1.30 (0.56) | 1.30 (0.39)
  42 months: number analyzed (Participants) | 15 | 18
  42 months | 1.43 (0.58) | 1.50 (0.49)
  54 months: number analyzed (Participants) | 15 | 16
  54 months | 1.58 (0.70) | 1.45 (0.50)

8. Secondary Outcome: AUC C-peptide From OGTT Over Time
Description: OGTT is performed at baseline, after 6 months and thereafter annually
Time Frame: During 5 year follow-up from treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nmol*min/L
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Number analyzed (Participants) | 24 | 24
nmol*min/L
  0 months | 134.82 (55.36) | 146.98 (62.12)
  6 months: number analyzed (Participants) | 23 | 24
  6 months | 121.07 (34.37) | 149.01 (54.66)
  18 months: number analyzed (Participants) | 20 | 20
  18 months | 149.88 (47.40) | 152.02 (52.66)
  30 months: number analyzed (Participants) | 21 | 18
  30 months | 157.35 (59.83) | 172.23 (50.24)
  42 months: number analyzed (Participants) | 12 | 15
  42 months | 169.48 (65.87) | 182.14 (76.33)
  54 months: number analyzed (Participants) | 15 | 16
  54 months | 183.23 (64.78) | 184.14 (65.59)

9. Secondary Outcome: HbA1c
Description: At all visits in the study HbA1c is measured. The change in HbA1c from baseline HbA1c is analysed at Laboratory of Clinical Chemistry, Skåne University Hospital, Malmö
Time Frame: During 5 year follow-up
Population: Children meeting the primary endpoint type 1 diabetes are not included in the analysis - therefore the number of analysed children drops during follow-up. Some data missing
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Number analyzed (Participants) | 25 | 25
mmol/mol
  0 months | 33.84 (3.52) | 32.76 (3.13)
  6 months | 34.88 (2.68) | 33.28 (2.92)
  12 months: number analyzed (Participants) | 24 | 25
  12 months | 34.92 (4.16) | 33.13 (3.0)
  18 months: number analyzed (Participants) | 24 | 22
  18 months | 36.63 (9.46) | 33.64 (3.36)
  24 months: number analyzed (Participants) | 21 | 22
  24 months | 34.14 (3.23) | 34.95 (6.09)
  30 months: number analyzed (Participants) | 21 | 20
  30 months | 35.19 (4.07) | 33.25 (2.81)
  36 months: number analyzed (Participants) | 18 | 19
  36 months | 33.94 (4.04) | 33.58 (4.34)
  42 months: number analyzed (Participants) | 16 | 18
  42 months | 33.19 (3.08) | 32.44 (3.03)
  48 months: number analyzed (Participants) | 15 | 18
  48 months | 32.40 (2.95) | 32.17 (2.62)
  54 months: number analyzed (Participants) | 15 | 16
  54 months | 33.73 (3.97) | 33.75 (2.74)
  60 months: number analyzed (Participants) | 16 | 16
  60 months | 34.56 (4.23) | 34 (3.12)

10. Secondary Outcome: First-phase Insulin Response From IvGTT Over Time
Description: As secondary variables of effect we will measure the change in first-phase insulin response. In all children a baseline IvGTT is performed and after that annual IvGTT´s are performed within the study. First phase insulin response is calculated from insulin 1 and 3 minutes after the given glucose solution. Insulin is measured by Laboratory of Clinical Chemistry at Skåne University Hospital, Malmö. Change in first phase insulin response will be calculated for each individual and compared between the groups.
Time Frame: During 5 year follow-up from treatment
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
Number analyzed (Participants) | 25 | 25
nmol/L
  0 months | 47.40 (42.42) | 55.52 (35.89)
  12 months: number analyzed (Participants) | 23 | 22
  12 months | 68.57 (54.17) | 66.00 (39.91)
  24 months: number analyzed (Participants) | 20 | 18
  24 months | 77.45 (61.36) | 70.27 (36.61)
  36 months: number analyzed (Participants) | 16 | 17
  36 months | 70.19 (38.55) | 81.06 (37.34)
  48 months: number analyzed (Participants) | 13 | 16
  48 months | 106.92 (66.97) | 84.75 (37.77)
  60 months: number analyzed (Participants) | 15 | 15
  60 months | 97.60 (63.15) | 89.60 (63.60)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were recorded during 5 year follow-up.
Arm/Group | Placebo Comparator | Alum-GAD (Diamyd)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25 | 2/25
Other Adverse Events (participants affected / at risk) | 25/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Comparator (N=25) | Alum-GAD (Diamyd) (N=25)
Pneumonia (Infections and infestations) | 1 | 0 — Inpatient warded pneumonia
arm fracture (Injury, poisoning and procedural complications) | 1 | 2 — In patient warded arm fractures after fall
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Comparator (N=25) | Alum-GAD (Diamyd) (N=25)
Ear pain (Ear and labyrinth disorders) | 2 | 0
Eye pruritus (Eye disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 6
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Tootache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 4
Fatigue (General disorders) | 0 | 2
Injection site reaction (General disorders) | 23 | 24
Malaise (General disorders) | 1 | 2
Pyrexia (General disorders) | 19 | 10
Celiac disease (Immune system disorders) | 2 | 2
Allergic conjunctivitis (Immune system disorders) | 1 | 0
Henoch Shoenlein Purpura (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 3
Seasonal allergy (Immune system disorders) | 2 | 3
Carbuncle (Infections and infestations) | 0 | 1
Chlamydia infection (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 4 | 0
Coxachie viral infection (Infections and infestations) | 1 | 0
Ear infection (Immune system disorders) | 6 | 3
Enterobiasis (Infections and infestations) | 2 | 2
Ebstein Barr Virus (Infections and infestations) | 0 | 1
Erythema Infectiosum (Infections and infestations) | 1 | 0
Gastoenteritis (Infections and infestations) | 17 | 19
Impetigo (Infections and infestations) | 1 | 0
Infected bite (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 4 | 7
Nasopharyngitis (Infections and infestations) | 21 | 21
Otitis externa (Infections and infestations) | 2 | 0
Otitis media (Infections and infestations) | 3 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2
Pseudocroup (Infections and infestations) | 0 | 1
Scarlet fever (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 1

LIMITATIONS AND CAVEATS:
Limitations: This study was a first study of Alum-GAD in non-diabetic children with multiple islet autoantibodies. The study was small in sample size which may limit the power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No